CLINICAL TRIAL: NCT05547490
Title: Treatment Patterns, Clinical Outcomes and Healthcare Resource Utilization Among Adult Patients With Moderate-To-Severe Plaque Psoriasis in Real-World Settings in China
Brief Title: A Study to Assess Treatment Patterns, Clinical Outcomes and Healthcare Resource Utilization Among Adult Participants With Moderate-To-Severe Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-206
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis
Keywords: Moderate to Severe Plaque PsO
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate-to-severe Plaque PsO: Participants experiencing moderate-to-severe plaque PsO, who have had at least one clinical visit.

SUMMARY:
The purpose of this study is to achieve a better understanding of clinical characteristics, treatment patterns and clinical outcomes of participants with moderate-to-severe plaque psoriasis (PsO) as well as their unmet medical needs and disease burden in real-world setting in China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-to-severe plaque PsO either confirmed by a dermatologist or meeting criteria of: BSA ≥ 3% or PASI ≥ 3 or Dermatology Life Quality Index (DLQI) ≥ 6.

Exclusion Criteria:

* Participating in Randomized controlled trial (RCT) between 1st January 2018 and 31st December 2021, if there was any.
* Diagnosis of erythrodermic psoriasis, pustular psoriasis or guttate psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants experiencing moderate-to-severe plaque PsO, who have at least one clinical visit (either outpatient or inpatient visit) between 1st January 2018 and 31st December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 3506 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Distribution of demographic characteristics: Age | Baseline
Distribution of demographic characteristics: Sex | Baseline
Distribution of clinical characteristics: Height | Baseline
Distribution of clinical characteristics: Weight | Baseline
Distribution of clinical characteristics: Body Mass Index (BMI) | Baseline
Distribution of clinical characteristics: Disease duration | Baseline
Distribution of clinical characteristics: Severity of PsO | Baseline
Distribution of clinical characteristics: Comorbidities | Baseline
Treatment patterns: Drug categories treated during study period | Up to 4 Years
Treatment patterns: Drug names treated during study period | Up to 4 Years
Treatment patterns: Medication dosage | Up to 4 Years
Treatment patterns: Drug's administration frequency | Up to 4 Years
Treatment patterns: Reason for treatment change during study period | Up to 4 Years
Treatment patterns: Treatment duration of each drug during study period | Up to 4 Years
Treatment patterns: Treatment sequence | Up to 4 Years
Treatment patterns: Change of treatment pattern | Up to 4 Years

SECONDARY OUTCOMES:
Number of participants achieving Body Surface Area of <3% during study period | Up to 4 Years
Psoriasis Area and Severity (PASI) Index | Up to 4 Years
Number of participants achieving Static Physicians Global Assessment (sPGA) of 0/1 during study period | Up to 4 Years
Healthcare resource utilization (HCRU) | Up to 4 Years
  HCRU will include visit date, visit type, cost, inpatient visits, outpatient visits, length of stay, and direct medical cost.
Evaluation of patient reported outcome measure: Patients' global assessment of disease activity (PtGA) | Up to 4 Years
  PtGA of psoriasis is an indicator of disease severity of PsO measured using a single-item, five- point scale ranging from 0 (clear) to 4 (severe). Category labels include 'clear', 'almost clear', 'mild', 'moderate' and 'severe'.
Evaluation of patient reported outcome measure: Dermatology life quality index (DLQI) | Up to 4 Years
  DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult participants with skin diseases such as eczema, psoriasis, acne and viral warts. Each item has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30 and higher scores indicate greater HRQoL impairment.
Evaluation of patient reported outcome measure: EQ-5D-3L | Up to 4 Years
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each dimension, participant is asked to choose one of the 3 levels (no problems, some problems, and extreme problems) to indicate his/her health state. This decision results into a 1-digit number and the digits for the five dimensions can be combined into a 5-digit number that describes the participant's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution - 0002, Beijing, Beijing Municipality
  - Local Institution - 0001, Nanjing, Jiangsu

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html